CLINICAL TRIAL: NCT05706038
Title: Impact of Adalimumab Withdrawal or Continuation on Severity of COVID-19 and Risk of IMID Relapse
Acronym: COV-ADA
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Gastroenterologist, IRCCS San Raffaele
Other Study IDs: COV-ADA
Record Dates: First submitted 2023-01-30; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Diseases; Rheumatic Disorder
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Adalimumab — Adalimumab is a fully human, high-affinity, recombinant anti-tumor necrosis factor (TNF) alpha monoclonal antibody used to treat rheumatoid arthritis, ankylosing spondylitis, psoriasis, psoriatic arthritis, Crohn disease, ulcerative colitis, etc.
  Adalimumab is a fully human, high-affinity, recombinant immunoglobulin G (IgG) anti-TNF alpha monoclonal antibody. It is a molecule comprising 1330 amino acids and has a molecular weight of approximately 148 kDa.[4] It inhibits the binding of TNF alpha (both soluble and membrane-bound) to its receptor. Specifically, it inhibits TNF alpha's interaction with p55 (TNFR1) and p75 (TNFR2) cell surface TNF receptors, which in turn interferes with cytokine-driven inflammatory processes. It is identical in structure and function to the naturally occurring human IgG1 and thus has high selectivity for TNF alpha and has low immunogenic potential.

SUMMARY:
This study is a retrospective pharmacological study, of a historical cohort. Collection of Retrospective data from February 2020 to 30 September 2021 The index date is the date of COVID-19 positive PCR test. The data will be collected until last news (last clinical visit or death).

There are no defined study visits. In the course of the study, the clinical data recorded are those corresponding to the standard medical procedure.

The goal of this study is to assess the impact on continuing or stopping adalimumab treatment on the occurrence of a severe COVID-19 (Coronavirus Disease 2019) in patients with Immune-Mediated Inflammatory Disease (IMID), during the first month after the diagnosis of SARS-CoV-2 infection.

To our knowledge, no comparisons have been performed between IMID patients stopping or not their maintenance treatment. In the context of the COVID-19 epidemic, the goal is to minimize the risk of disease flare while simultaneously minimizing the risk of severe COVID-19. In this study, we hypothesized that patients treated by adalimumab for IMID might not be susceptible to severe COVID-19 disease course.

DETAILED DESCRIPTION:
Immune-mediated inflammatory disease (IBD or rheumatic disease) patients treated with adalimumab with positive PCR COVID-19 diagnosis will be enrolled by physicians.

There will be four predefined and balanced group:

1. Adalimumab withdrawal in patients with IBD
2. Adalimumab continuation in patients with IBD
3. Adalimumab withdrawal in patients with RA, PsA, axSpA, and nrxSpA
4. Adalimumab continuation in patients with RA, PsA, axSpA, and nrxSpA n = 312 subjects for groups 1+3 together and 312 subjects for groups 2+4 together.

All data will be described by percentages (categorical variables) and mean +/- standard deviation and quartiles (continuous variables). The median time of follow-up survival data will also be detailed for each event of interest (admission to intensive care unit, need to a mechanical ventilation during hospitalization, death). Kaplan Meier curve will describe the probability of the occurrence of a severe SARS-CoV-2 infection (see primary endpoint for definition).

Time to analysis - better define - time to severity of the event. Occurrence (yes/no)

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years
2. diagnosis of immune-mediated inflammatory disease:

   1. IBD: CD, UC or undetermined colitis
   2. Rheumatic diseases: RA, PsA, axSpA, and nrx SpA
3. patients treated with adalimumab for IMID at time of SARS-CoV-2 infection diagnosis
4. COVID-19 positive PCR test
5. minimum treatment duration on adalimumab of 3 months before SARS-CoV-2 infection diagnosis
6. minimum follow-up of one month after SARS-CoV-2 infection diagnosis

Exclusion Criteria:

1. Adalimumab withdrawal for other reasons than SARS-CoV-2 infection
2. Patients with COPD or lung co-morbidities
3. Pregnant, parturient, or breastfeeding woman
4. Minor person (non-emancipated)
5. Adult person under legal protection (any form of public guardianship)
6. Adult person incapable of giving consent and not under legal protection
7. Person deprived of liberty for judicial or administrative decision, person under psychiatric care as referred in articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective pharmacological study of a historical cohort: retrospective data from February 2020 to September 2021.
  Immune-mediated inflammatory disease (IBD or rheumatic disease) patients treated with adalimumab with positive Polymerase Chain Reaction (PCR) COVID-19 diagnosis.
  624 patients will be needed (of whom 312 with maintenance of treatment).
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
composite endpoint: occurrence of an admission to intensive care unit and/or need to a mechanical ventilation during hospitalization and/or death | first month after the diagnosis of SARS-CoV-2 infection
  The primary endpoint is the occurrence of a severe SARS-CoV-2 infection, which will be defined by a composite endpoint: occurrence of an admission to intensive care unit and/or need to a mechanical ventilation during hospitalization and/or death, during the first month after the diagnosis of SARS-CoV-2 infection.

SECONDARY OUTCOMES:
occurrence of IMID flare | from diagnosis of SARS-CoV-2 infection to enrollment
  to measure the occurrence of IMID flare, which will be assessed by the occurrence of a disease flare until last clinical visit, to evaluate risk factors for severe COVID-19, and to evaluate risk factors for IMID flare. IMID flare is defined by patient requiring medical intervention (additional treatment and/or dose escalation and/or surgery and/or hospitalization).

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Irccs Ospedale San Raffaele, Milan, Italy